CLINICAL TRIAL: NCT07013578
Title: A Randomized Evaluation of Changes in Anxiety and Depression in Inflammatory Bowel Disease Patients Comparing Structured Mental Health Support to App Based Mental Health Support in Addition to Standard of Care Medical Treatment
Brief Title: TIDHI Mental Health in IBD Patients Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TIDHI Innovation Inc. (Other)
Collaborators: Amgen (Industry); Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3665
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD)
Keywords: Healing Circuits
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sessions with a social worker based on Healing Circuits™ Methodology (Experimental)
  Interventions: Behavioral: Healing Circuits™ sessions
- Online modules of a self-directed Healing Circuits™ curriculum (Experimental)
  Interventions: Behavioral: self-directed Healing Circuits™ curriculum

INTERVENTIONS:
Behavioral: Healing Circuits™ sessions — Treatment of the Study group will involve 12-weekly 50-minute sessions with a social worker who has been trained in the Healing Circuits™ Methodology - a structured mental health support delivered by a therapist in a one-on-one model.
  Arms: Sessions with a social worker based on Healing Circuits™ Methodology
Behavioral: self-directed Healing Circuits™ curriculum — Treatment of the Control group will involve 12 weekly online modules of a self-directed Healing Circuits™ curriculum - structured mental health support being delivered in an web-based video instruction model.
  Arms: Online modules of a self-directed Healing Circuits™ curriculum

SUMMARY:
The purpose of this study is to test the impact of Healing Circuits™; a structured mental health support model on IBD patients. The eligible study participants will be randomly divided into two groups: 1. the group receiving structured mental health support with a social worker and 2. the group receiving structured mental health support via a self-directed online curriculum. Both groups will be receiving the same type of therapy, Healing Circuits™, but the group receiving the therapy via the online self-directed curriculum will be receiving the therapy mostly by web-based video instruction. The two groups will be evaluated over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet each of the following criteria for enrolment into the study:

1. Written informed consent must be obtained and documented.
2. Males and females between the ages of 18 and 75 years of age with documented diagnosis of IBD.
3. GAD7 and/or PHQ9 score of 10 - 15.
4. Ability of subject to participate fully in all aspects of this clinical trial.
5. IBD patients who plan to have ongoing medical care at TIDHI.

Exclusion Criteria:

Subjects who exhibit any of the following conditions are to be excluded from the study:

1. Plan for change in systemically delivered IBD-related medical therapy in the 3 months after screening.
2. Serious underlying psychiatric disorder such as schizophrenia or bipolar disorder.
3. Planned change in psychiatric medication, if any is being taken, within 3 months after screening.
4. History of illegal drug abuse (excluding marijuana) or alcohol abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder 7-item Scale (GAD-7) Score | 3 months following initiation of Healing Circuits™
  The Generalized Anxiety Disorder Assessment (GAD7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Scores range from 0 to 21, with higher scores indicating greater anxiety.
  This outcome will compare the mean change in GAD-7 scores from baseline between participants receiving one-on-one therapy and those receiving app-based therapy.
Time to Improvement in Generalized Anxiety Disorder 7-item Scale (GAD-7) Score | 3 months following initiation of Healing Circuits™
  Improvement is defined as a ≥2-point reduction from baseline in GAD-7 score. The outcome will compare the time (months ) it takes participants in the one-on-one therapy group and the app-based therapy group to reach this level of improvement.
Change in Patient Health Questionnaire-9 (PHQ-9) Score | 3 months following initiation of Healing Circuits™
  PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Scores range from 0 to 27, with higher scores indicating greater depression severity.
  This outcome will assess the mean difference in PHQ-9 scores between the one-on-one therapy and app-based therapy groups.
Time to Improvement in Patient Health Questionnaire-9 (PHQ-9) Score | 3 months following initiation of Healing Circuits™
  Improvement is defined as a ≥2-point reduction from baseline in PHQ-9 score. This outcome compares the time (months ) it takes for participants in the one-on-one therapy group and the app-based therapy group to reach the improvement threshold.

SECONDARY OUTCOMES:
Proportion of Participants Achieving at Least a 2-Point Reduction in GAD-7 Score | 6, 9, and 12 months following initiation of Healing Circuits™
  This outcome measures the proportion of participants who experience a reduction of at least 2 points in the GAD-7 (range: 0-21, higher scores = worse anxiety) at 6, 9, and 12 months after beginning the Healing Circuits™ intervention.
Proportion of Participants Achieving at Least a 2-Point Reduction in PHQ-9 Score | This outcome measures the proportion of participants who experience a reduction of at least 2 points in the PHQ-9 (range: 0-27, higher scores = worse depression) at 6, 9, and 12 months after beginning the Healing Circuits™ intervention.
  6, 9, and 12 months following initiation of Healing Circuits™
Mean Change in 36-Item Short Form Survey (SF-36) Score Between Groups | 3, 6, 9, and 12 months following initiation of Healing Circuits™
  This outcome measures the mean difference in scores on the SF-36, a 36-item, patient-reported survey of patient health. Each item is scored out of 100 and a higher score is correlated to more favorable health. It addresses 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  The comparison will be made between the one-on-one therapy group and the app-based therapy group at the specified time points.
Mean Change in Patient Satisfaction Score on a Likert Scale Between Groups | 3, 6, 9, and 12 months following initiation of Healing Circuits™
  This outcome measures the mean difference in patient satisfaction between the one-on-one therapy group and the app-based therapy group. Satisfaction is assessed using a custom 10-point Likert scale ranging from 1 (Worst Possible Experience) to 10 (Best Possible Experience), with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Silverberg, MD, PhD, Principal Investigator — TIDHI Innovation Inc.; Marci Reiss, DSW, Principal Investigator — TIDHI Innovation Inc.
Locations (1):
- Toronto Immune and Digestive Health Institute, North York, Ontario, Canada